CLINICAL TRIAL: NCT02046278
Title: LifeSeal™ Pilot Study in Subjects Undergoing Circular Stapled Anastomosis Created Within 10 cm of the Anal Verge
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LifeBond Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLP-LS-0110
Record Dates: First submitted 2014-01-23; First posted 2014-01-27 (Estimated); Last update posted 2016-08-30 (Estimated); Status verified 2016-08

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control arm - Standard of Care (No Intervention): The anastomosis will be created using Standard of Care only
- Device arm - Standard of Care + LifeSeal™ Kit (Experimental): The anastomosis will be created using SOC + LifeSeal™ Kit
  Interventions: Device: LifeSeal™ Kit

INTERVENTIONS:
Device: LifeSeal™ Kit
  Arms: Device arm - Standard of Care + LifeSeal™ Kit

SUMMARY:
A Pilot Study in Subjects Undergoing circular stapled anastomosis created within 10 cm of the anal verge.

ELIGIBILITY:
Inclusion Criteria:

1. Subject, or authorized representative, signed a written Informed Consent Form
2. Subject is 18 years or older
3. Subject is scheduled for elective open or laparoscopic surgery involving the creation of a circular stapled anastomosis created within 10cm from the anal verge.
4. If female - not be of child bearing potential, or be using acceptable contraception methods.
5. Subject participating in studies involving approved drug or device will be enrolled only following a mutual consideration of the investigator together with the Sponsor.

Exclusion Criteria:

1. Subject has a history of hypersensitivity to porcine derived gelatin or collagen
2. Subject participating in any other study involving an investigational (unapproved) drug or device.
3. Subject with a BMI higher than 40
4. Female Subject states that she is pregnant or breast feeding
5. Subject with ASA status higher than 3
6. Avastin use within 30 days prior to surgery
7. Subject who underwent a prior pelvic anastomosis
8. Subject is scheduled for another surgery during the follow up period of this study (not including stoma closure)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2014-01; Primary Completion 2014-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Assessment of the overall Subject safety by incidence of pre specified procedure related Adverse Events. | Up to 15 weeks

SECONDARY OUTCOMES:
Performance Rate of anastomotic leak (both radiological and clinical leaks) | Up to 15 weeks post procedure or at stoma closure, whichever comes first

CONTACTS AND LOCATIONS:
Locations (8):
- Belgium (4):
  - OLV Ziekenhuis, Aalst
  - Ziekenhuis Oost-Limburg, Genk
  - University Hospital, Ghent
  - UZ Leuven, Leuven
- Sourasky Medical Center, Tel Aviv, Israel
- Sweden (3):
  - Skane University Hospital, Malmo
  - Karolinska Institutet, Stockholm
  - Uppsala University Hospital, Uppsala